CLINICAL TRIAL: NCT00291356
Title: A Double-blind, Randomized, Placebo-controlled, Repeat Dose Study to Compare the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK189075 With GW869682 in Subjects With Type 2 Diabetes Mellitus
Brief Title: GSK189075, GW869682 Or Placebo In Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: KG2104940
Record Dates: First submitted 2006-02-13; First posted 2006-02-14 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Diabetes Mellitus, Type 2; Non-Insulin-Dependent Diabetes Mellitus
Keywords: Diabetes; sodium dependent glucose transporter; SGLT2; GSK189075; GSK189074; SGLT1; GW869683
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

INTERVENTIONS:
Drug: GSK189075 oral tablets
Drug: GW869682 oral tablets
  Other Names: GSK189075 oral tablets

SUMMARY:
This is a study to compare the safety, blood concentrations, and effects of GSK189075, GW869682, and placebo when dosed for 2-weeks by mouth to patients with type 2 diabetes.

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes.
* HbA1c (a measure of the average amount of sugar in blood over the last 2 or 3 months) levels are between 7.0 and 9.0.
* Taking 850mg or more per day metformin, but not taking any other diabetes medications.
* Must be medically able and willing to discontinue diabetic medications from at least 2 weeks prior to first study dose until the last study assessment.
* Diabetic subjects who have not yet started taking diabetes medications or whose diabetes is controlled by diet alone may also be eligible to enroll if their HbA1c is within 7.5 to 9.0.
* Women may be eligible if they are post-menopausal or surgically sterile.
* If taking ACE inhibitors, beta-blockers, calcium channel blockers, or statin type drugs, you may be eligible if your dose has been stable for at least 30 days prior to the start of the clinical trial.

Exclusion criteria:

* Using illicit drugs, or have antibodies to hepatitis B, hepatitis C, or HIV.
* Have any major health problems other than type 2 diabetes.
* Require insulin therapy or oral antidiabetic medication other than metformin.
* Subjects who have had a urinary tract infection within 4 weeks of the start of the study or who have kidney disease.
* Subjects with either low or high blood pressure.
* Men who are unwilling to abstain from intercourse, or use a condom with a pregnant or nursing female, or who are unwilling to use a condom with another form of contraception with a female who could become pregnant.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: side effects and relevant changes in blood pressure, heart rate and ECG measurements, blood and urine measurements, the amount of fluid taken in and excreted, and kidney function will be monitored over course of study.

SECONDARY OUTCOMES:
Amount and percentage of glucose excreted in urine by kidneys. Effect of compounds on lipid metabolism analysed.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Chula Vista, California, United States
- Germany (2):
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Berlin, State of Berlin